CLINICAL TRIAL: NCT06757400
Title: Τhe Effect of Lumbar Spine Mobilization and Manipulation on Pressure Pain Threshold in Patients with Non-specific Chronic Low Back Pain: a Cross-over Randomised Controlled Trial
Brief Title: Τhe Effect of Lumbar Spine Mobilization and Manipulation on Pressure Pain Threshold in Patients with NSLBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of West Attica (Other)
Responsible Party: Principal Investigator, Stefanos Karanasios, Associate Professor, Physiotherapy Dept, University of West Attica, University of West Attica
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 65273- 07/07/2023
Record Dates: First submitted 2024-05-26; First posted 2025-01-03 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Low Back Pain; Lumbago
Keywords: non-specific low back pain; manual therapy; hypoalgesia; pressure pain threshold
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mobilization (Experimental): 27 patients with chronic low back pain will be assigned to receive one intervention with grade IV posteroanterior (PA) mobilization in the Lumbar spine
  Interventions: Other: Mobilization; Other: manipulation
- Manipulation (Active Comparator): 27 patients with chronic low back pain will be assigned to receive one intervention with lumbar manipulation
  Interventions: Other: Mobilization; Other: manipulation

INTERVENTIONS:
Other: Mobilization — Mobilization will be conducted on an examination table with the subject in prone position. Therapist will place his hypothenar to the most hypomobile lumbar spine segment after assessment.It will be a posteroanterior (PA) direction tecnique, Maitland's GRADE 4, 3 sets of 60 seconds duration for each set.
Other: manipulation — Manipulation will be conducted on an examination table with the subject in right lateral decubitus. It will be a rotary manipulation to the most hypomobile lumbar spine segment after assessment.

SUMMARY:
Manual therapy, including mobilizations and manipulations, appears to be as effective as other types of therapy for chronic low back pain.

The aim of this cross-sectional study is to compare the effects of lumbar spine mobilization and manipulation on the pressure pain threshold in patients with non-specific chronic low back pain.

DETAILED DESCRIPTION:
Background: Manual therapy, including mobilizations and manipulations, appears to be equally effective as other types of therapy for chronic low back pain. According to the Orthopaedic Section of the American Physical Therapy Association (APTA), there is evidence indicating that these techniques can reduce pain, improve spinal and hip mobility, and decrease disability in patients with low back pain. The aim of this study is to compare the effects of lumbar spine mobilization and manipulation on the pressure pain threshold in patients with non-specific chronic low back pain.

Methods: The present study will be a cross-sectional study in which participants will be men and women aged 18 to 60 years. The sample size was estimated by effect size, with a minimum of 27 participants required to provide statistically or clinically significant results. Each subject will receive two interventions-mobilization or manipulation-on two different days, in a random order. The primary outcomes will be pain perception, including subjective pain intensity and pressure pain threshold. Secondary outcomes will include the range of motion (ROM) of lumbar spine flexion, extension, and lateral flexion. Data will be collected before and after each intervention. Assessors will use a digital algometer, an electronic inclinometer, and a numerical rating scale (NRS). ANOVA and t-test calculations will be performed on data processed by SPSS Version 25 to analyze results for all outcomes. The level of significance will be set at 5% (p = 0.05) with a confidence interval of 95% (CI = 95%).

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 years old
* diagniosed with non specific low back pain
* symptoms lasting for more than 12 weeks

Exclusion Criteria:

* spinal fractures,
* neurological impairment due to herniated spinal disc,
* spondylolisthesis,
* joint degenerative diseases,
* osteoporosis,
* spinal infections,
* cauda equina syndrome,
* spinal tumors or bone marrow malignancies,
* spinal surgeries
* history of cancer,
* use of steroids

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2023-11-04 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
1. Pressure pain threshold | Baseline and 15 minutes
  Changes between pre- and post- intervention in Pressure Pain Threshold will be measured using at the L5 spinous process, upper trapezius muscle the tibialis anterior muscle. The COMPACT DIGITAL ALGOMETER CAPACITIES TO: 100 lbf / 50 kgf / 500 N, will be used by an independent assessor. The assessor will be blinded to participants' group.

SECONDARY OUTCOMES:
Range Of Motion (ROM) | Baseline and 15 minutes
  ROM will be measured in sagittal (flexion and extension) and frontal planes (right and left lateral bending) using an electronic goniometer. The participants will perform each movement three times were performed and the average will be recorded for the analysis
Pain Intensity | Baseline and 15 minutes
  Participants will complete a self- reported numerical pain rating scale (NRS) from 0-10, with "0" indicated no pain and "10" the maximum possible pain, covering pain intensity over the past week

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Sampsonis, Peristeri, Αττικης, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dal Farra F, Risio RG, Vismara L, Bergna A. Effectiveness of osteopathic interventions in chronic non-specific low back pain: A systematic review and meta-analysis. Complement Ther Med. 2021 Jan;56:102616. doi: 10.1016/j.ctim.2020.102616. Epub 2020 Nov 13. PMID 33197571
- [Background] Childs JD, Fritz JM, Flynn TW, Irrgang JJ, Johnson KK, Majkowski GR, Delitto A. A clinical prediction rule to identify patients with low back pain most likely to benefit from spinal manipulation: a validation study. Ann Intern Med. 2004 Dec 21;141(12):920-8. doi: 10.7326/0003-4819-141-12-200412210-00008. PMID 15611489
- [Background] Rubinstein SM, de Zoete A, van Middelkoop M, Assendelft WJJ, de Boer MR, van Tulder MW. Benefits and harms of spinal manipulative therapy for the treatment of chronic low back pain: systematic review and meta-analysis of randomised controlled trials. BMJ. 2019 Mar 13;364:l689. doi: 10.1136/bmj.l689. PMID 30867144
- [Background] Arribas-Romano A, Fernandez-Carnero J, Molina-Rueda F, Angulo-Diaz-Parreno S, Navarro-Santana MJ. Efficacy of Physical Therapy on Nociceptive Pain Processing Alterations in Patients with Chronic Musculoskeletal Pain: A Systematic Review and Meta-analysis. Pain Med. 2020 Oct 1;21(10):2502-2517. doi: 10.1093/pm/pnz366. PMID 32100027
- [Background] Coronado RA, Gay CW, Bialosky JE, Carnaby GD, Bishop MD, George SZ. Changes in pain sensitivity following spinal manipulation: a systematic review and meta-analysis. J Electromyogr Kinesiol. 2012 Oct;22(5):752-67. doi: 10.1016/j.jelekin.2011.12.013. Epub 2012 Jan 30. PMID 22296867